CLINICAL TRIAL: NCT00720122
Title: Effects of Recombinant Human Insulin Like Growth Factor-1 (rhIGF-1) on Bone Metabolism in Adolescent Girls With Anorexia Nervosa
Brief Title: Effects of rhIGF-1 on Bone Metabolism in Adolescent Girls With Anorexia Nervosa
Acronym: 814
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Asssociate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MassGH; CDER
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Disorder of Bone Density and Structure, Unspecified
Keywords: Bone density; Bone turnover markers; rhIGF-1; Bone structure; Anorexia nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anorexia Nervosa Females (Experimental)
  Interventions: Drug: Recombinant human insulin like growth factor-1 (rhIGF-1)

INTERVENTIONS:
Drug: Recombinant human insulin like growth factor-1 (rhIGF-1) — Twice daily
  Other Names: Tercica

SUMMARY:
Adolescents and young adults with anorexia nervosa (AN) are at high risk for low bone mineral density at a time when healthy adolescents are rapidly accruing bone, with implications for peak bone mass and fracture risk in later life. They are also deficient in insulin-like growth factor 1 (IGF-1), the bone trophic factor made in the liver in response to growth hormone (GH), despite elevated levels of growth hormone. It is possible that deficiency of insulin-like growth factor 1, a hormone very important for the maintenance of skeletal integrity, may contribute to the severe osteopenia seen in anorexia nervosa. The physiologic effects of recombinant human insulin-like growth factor 1 (rhIGF-1) treatment in adolescents and young adults with anorexia nervosa have not been studied. The goal of this proposal is to investigate the effects of recombinant human insulin-like growth factor 1 on bone density and bone microarchitecture in adolescent girls and young adult women with anorexia nervosa over a 6 month period. We hypothesize that adolescent and young adult anorexia nervosa patients, being insulin-like growth factor 1 deficient, will respond to exogenously administered recombinant human insulin-like growth factor 1 with elevations in biochemical indices of bone turnover and an increase in bone density and improvement in bone structure, or maintain bone density (in contrast to the decrease in bone density expected in adolescent girls and women with anorexia nervosa who are not treated).

ELIGIBILITY:
Inclusion Criteria:

- Meet criteria for anorexia nervosa (AN) as described in the Diagnostic and Statistical Manual of Mental Disorders

Exclusion Criteria:

* Pregnant or nursing
* Hematocrit < 30%, K < 3 mmol/L
* Any illness (other than AN) known to affect bone and mineral metabolism such as diabetes, untreated hypo- or hyperthyroidism, or hyperparathyroidism
* History of use of any medicine, such as corticosteroids, known to affect bone density. Subjects who are on estrogen will still be eligible to participate in the study because our data in adult women with AN do not indicate deleterious effects of estrogen in patients receiving rhIGF-

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, Principal Investigator — MD
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anorexia Nervosa Females: Females aged 12 - 26 years Subjects received 30 mcg/kg/dose of recombinant human insulin like growth factor-1 (rhIGF-1) twice daily subcutaneously
Period: Overall Study
Arm/Group | Anorexia Nervosa Females
Started | 28
Completed | 19
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Anorexia Nervosa Females
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.142857 (3.6180032)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Spine Bone Density (g/cm^2)
Description: Change in spine bone density over 6 months (6month data- baseline data). Bone density at the spine was assessed using dual energy x-ray absorptiometry at baseline and 6 months and the change in bone density over these 6 months was calculated.
Time Frame: Baseline and 6 months
Population: The study participants analyzed were those that completed the first 6 months of the study and had a bone density performed at the baseline visit and then again at the 6 month visit as per protocol.
Measure: Mean (Standard Error); unit: gm/cm^2
Arm/Group | Anorexia Nervosa Females
Number analyzed (Participants) | 19
gm/cm^2 | -0.00558 (0.00653)
Statistical Analysis 1: Comparison: Anorexia Nervosa Females; A paired t-test was performed. The null hypothesis was that bone density would decrease over 6 months in females with anorexia nervosa, as observed in life course studies; Test type: Superiority or Other; p = 0.40, Paired t-test; Mean Difference (Final Values) = -0.00558, 95% CI 2-sided [-0.0081 to 0.0193], Standard Error of Mean 0.00653

ADVERSE EVENTS:
Time Frame: For the adolescent arm, adverse event data was collected for 6 months. For the adult arm, adverse event data was collected for 1 year.
Description: All subjects were assessed for any adverse events at screen, baseline, 1 month, 3 months, 4.5 months, and 6 months. The adult arm was subsequently assessed for any adverse events at 7 months, 9 months, and 12 months.
Arm/Group | Anorexia Nervosa Females
Serious Adverse Events (participants affected / at risk) | 5/28
Other Adverse Events (participants affected / at risk) | 22/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anorexia Nervosa Females (N=28)
Hospitalization (General disorders) | 4 (8) — These are unrelated and expected Serious Adverse Events and are due to the subjects' eating disorders.
Self-Injury (General disorders) | 1 (1) — This is an unrelated and expected Serious Adverse Event and is due to this subject's eating disorder and depression.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anorexia Nervosa Females (N=28)
Itchiness at Injection Site (General disorders) | 4 (6)
Facial Discoloration (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fall (General disorders) | 1 (1) — Subject fell while running for bus and suffered abrasions on left knee, shin, foot and hand.
Food Poisoning (Gastrointestinal disorders) | 1 (1) — Subject ate hummus and felt ill afterwards.
Elevated Aspartate Aminotransferase (General disorders) | 4 (9)
Severe Weight Loss (General disorders) | 1 (1) — Subject exhibited severe weight loss at 9 month study visit and was discontinued from study due to refusal of inpatient treatment, for safety reasons.
Vomiting (Gastrointestinal disorders) | 1 (1) — Subject stated it could be due to fatty food recently eaten.
Femoral Lymph Node Enlargement (General disorders) | 1 (1) — Subject reported this, but enlargement was not found on exam by study nurse practitioner.
Bruising (General disorders) | 4 (4) — One subject said this was due to her eating disorder and did not occur specifically at the injection site.
Cold with Mild Nose Bleed (General disorders) | 1 (1)
Lightheaded and Pale at Blood Draw (General disorders) | 1 (2)
Low Glucose Level (General disorders) | 1 (2)
Elevated Alanine Aminotransferase (General disorders) | 2 (2)
Heartburn (General disorders) | 2 (2) — One subject said that this was due to her calcium supplements.
Achiness (General disorders) | 1 (1)
Spider Bite (General disorders) | 1 (1)
Mild Itchiness to Bilateral Lower Extremities (General disorders) | 1 (1) — The subject stated that this was most likely due to her recent change in soap powder.
Breast Bone Pain (General disorders) | 1 (1) — The subject reported the pain lasting 5 -6 seconds and then resolving spontaneously.
Dizziness (General disorders) | 2 (2) — Coincided with the subject's recent Lexapro dose reduction.
Soreness at Injection Site (General disorders) | 1 (1)
Low Potassium Level (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (1)
Increased Fatigue (General disorders) | 1 (1) — Coincided with subject's increase in Prozac dosage.
Irritation at Injection Site (General disorders) | 8 (11)
Papules at Injection Site (General disorders) | 1 (1)
Abdominal Bloating (General disorders) | 1 (1)
Burning Sensation at Injection Site (General disorders) | 1 (1)
Poison Ivy Rash (General disorders) | 1 (1)
Prominent Thyroid (General disorders) | 1 (1) — The subject did not have a goiter. Her thyroid stimulating hormone, thyroxine, and triiodothyronine labs were all normal.
Swelling of Bilateral Feet (General disorders) | 1 (1) — Subject stated that this was probably due to warm weather.
Night Sweats (General disorders) | 1 (1) — Subject stated that this was mostly likely due to warmer weather and the temperature being higher in her apartment building.
Back Pain (General disorders) | 1 (1) — Subject had an ongoing history of back pain.
Joint Pain (General disorders) | 1 (1) — In subject's hand.
Hip Pain (General disorders) | 1 (1)
Headaches (General disorders) | 1 (1) — The subject had an ongoing history of headaches.
Erythema at Injection Site (General disorders) | 4 (4)
Elevated Insulin-like Growth Factor 1 (General disorders) | 1 (1)
Elevated Potassium Level (General disorders) | 1 (1)
Extremity Pain (General disorders) | 1 (1) — Subject felt pain in hand and wrist after school and occasionally during school.
Occasional Bleeding at Injection Site (General disorders) | 1 (1)
Kidney Stone (Renal and urinary disorders) | 1 (1) — Subject had a kidney stone that pass and was not tested. Subject followed up with a specialist and stopped taking calcium supplements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No